CLINICAL TRIAL: NCT01423214
Title: A Trial to Assess Robot-assisted Surgery and Laparoscopy-assisted Surgery in Patients With Mid or Low Rectal Cancer
Acronym: COLRAR
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Gyu-Seog Choi, Colorectal Cancer Center, Kyungpook National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KNUHCRC003
Record Dates: First submitted 2011-08-01; First posted 2011-08-25 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Rectal Cancer
Keywords: rectal cancer; robot; laparoscopy; total mesorectal excision; robotic surgery
MeSH Terms: conditions — Rectal Neoplasms | interventions — Robotic Surgical Procedures; Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Robotic LAR (Experimental): Individuals who underwent robot-assisted surgery for primary rectal cancer
  Interventions: Procedure: robot-assisted surgery
- Lap LAR (Active Comparator): Individuals who underwent laparoscopic surgery for primary rectal cancer
  Interventions: Procedure: Laparoscopic surgery

INTERVENTIONS:
Procedure: robot-assisted surgery — da Vinci surgical system® (Intuitive Surgical, Sunnyvale, CA, USA)
  Arms: Robotic LAR
Procedure: Laparoscopic surgery — Conventional laparoscopic procedures
  Arms: Lap LAR

SUMMARY:
This study sets up the final study end point and three detailed goals as the following.

The main objective of study: This trial is done to assess the safety and benefit of robotic resection compared with conventional laparoscopy-assisted resection for curative treatment of patients with cancer of the mid or low rectum.

Detailed goal of study:

The primary endpoint: This study is designed to assess whether robotic surgical system improves the quality of rectal cancer surgery, especially in total mesorectal excision quality and a circumferential margin positivity rate

The secondary endpoint: This study aims to compare 3- and 5-year disease-free survival and overall survival after robot and laparoscopic resection of distal rectal cancer. This study will also assess the pelvic autonomic nerve preservation, short-term morbidity, pathological quality (i.e. number of harvested lymph node), local recurrence, and blood loss during surgery.

DETAILED DESCRIPTION:
Recently, the efficacy and oncological safety of laparoscopy has been demonstrated for treating colon cancer, and similar long-term results at 5-year confirmed by the several multicenter study trial. However, conventional laparoscopic surgery for rectal cancer is technically more difficult than colonic resection because of the confined space in the pelvis and the limitations of existing laparoscopic instruments which have a restricted range of movement compared with the provided by the surgeon's hand. Consequently, recent studies which compared short-term outcomes between open and laparoscopic rectal resections have reported higher rates of conversion to open surgery, positive circumferential margins, and increased anastomotic leakage in patients who underwent laparoscopic approach.

The da Vinci® Surgical System (Intuitive surgical, Sunnyvale, CA, USA) was introduced as the next advance in minimally invasive surgery to overcome the technical limitations of laparoscopy. The advantages of robotic assistance include enhanced dexterity, improved three-dimensional vision, and more intuitive instrument manipulation. This device eases the technical challenges of the minimally invasive approach and may make a complex surgical task more accessible to surgeons without extensive laparoscopic experience.

With its dependence on precise dissection in a narrow pelvic cavity, it is anticipated that rectal cancer surgery is one of the indications most likely to benefit from robot assistance. However, it is difficult to conclude whether robot assistance leads to better outcomes because few studies have directly compared the three existing techniques. Although robotic rectal excision has been reported to be safe and feasible in the recent literatures, a number of these results were based on small number of case series. There have been no randomized trials demonstrating the safety of robotic surgery in the treatment of rectal cancer. This study is designed to assess the efficacy and safety of robotic surgery compared with that of laparoscopic surgery for mid or low rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility rule of enrollment
* Rectal adenocarcinoma that were 10 cm or less from the anal verge
* at least 18 years old & at most 80 years old
* Clinically diagnosed cT3N0-2 disease
* Clinical diagnosis of carcinoma involving a single rectal segment
* Patients with adequate hepatic, renal, and bone marrow function, and a left ventricular ejection fraction of 55% or higher measured by echocardiography

Exclusion Criteria:

* The presence of metastasis to the liver, lung, brain, bone, abdominal aortic lymph node, lateral pelvic wall lymph node and inguinal lymph node
* A past history of the cancer occurring in other body areas than the rectal cancer (except for a past history of the radical resection due to skin cancer)
* Severe cardiac diseases or failure
* Severe pulmonary diseases or dysfunction
* The presence of psychiatric diseases
* The concurrent presence of other severe medical diseases
* An ineligibility to participate in the clinical study based on the judgment of investigators from a legal perspective

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2013-06; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Surgical quality based on pathological examination | up to 4 weeks after operation
  A comparison of completeness of total mesorectal excision

SECONDARY OUTCOMES:
Postoperative morbidity | up to 30 dyas after operation
  A comparison of the postoperative recovery variables, the postoperative complications and mortality
Pelvic autonomic nerve preservation (intraoperative confirmation of pelvic nerve preservation) | The day of operation
  During procedure, a surgeon indentifies pelvic autonomic nerve and confirm whether the nerves are preserved or sacrificed.
Change from Baseline in QLQ 30, IIEF-5(5-item Version of the International Index of Erectile Function), IPSS(International Prostate Symptom Score), FSFI(Female Sexual Function Index), and Wexner's scoring | up to 12months after operation
  EORTC QLQ 30:an assessment tool for measuring the quality of life IIEF-5 : an assessment tool for measuring male erectile function IPSS : an assessment tool for measuring voiding function FSFI : an assessment tool for measuring female sexual function Wexner's scoring : an assessment tool for measuring anal sphincter function Time points : 1,3,6, and 12months after operation
5-year overall survival rate | up to 5 yearsa after operation
  A survival analysis will be performed using the Kaplan-Meier method, for which a comparison of the survival curve will also made using a Log-rank test.
5-year disease-free survival rate | up to 5 years after operation
  A survival analysis will be performed using the Kaplan-Meier method, for which a comparison of the survival curve will also made using a Log-rank test.

CONTACTS AND LOCATIONS:
Overall Officials: Gyu seog Choi, M.D, Study Chair — Kyunpook National Univercity Medical Center
Locations (3):
- South Korea (3):
  - Gyu seog Choi, Daegu
  - Nam Kyu Kim, Seoul
  - Seon-Hahn Kim, Seoul